CLINICAL TRIAL: NCT06260293
Title: The Effect of Post-operative Exercise in Gastric Cancer Patients: A Randomized Controlled Trial (RCT) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4-2022-0208
Record Dates: First submitted 2024-01-24; First posted 2024-02-15 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental)
  Interventions: Behavioral: exercise
- Usual care group (No Intervention)

INTERVENTIONS:
Behavioral: exercise — A total of 4 exercise interventions.
  Twice In-patient exercise interventions: exercises on the ward at POD1, and POD2, and Recommended walking and stretching.
  Twice home-based exercise interventions: post-discharge, Recommended 30 minutes of low to moderate-intensity walking and daily bodyweight exercises per day(150 minutes each week). and remote exercises 1 per week.
  Arms: Exercise group

SUMMARY:
Medical advancements are enhancing the survival rates of individuals with gastric cancer. The growing population of gastric cancer survivors underscores the importance of managing treatment-related after-effects and side effects. Diminished physical function in cancer patients, particularly following gastric cancer surgery, is linked to increased mortality. The substantial decline in physical activity post-surgery contributes to a notable reduction in cardiorespiratory fitness and lower extremity muscle strength. Early postoperative exercise has demonstrated positive outcomes in colorectal cancer patients, facilitating early hospital discharge and supporting long-term recovery. However, there is a paucity of research on the efficacy of early postoperative exercise in the context of gastric cancer. Therefore, this study aims to evaluate the impact of early postoperative exercise on physical function following gastric cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women 19 years of age or older
2. Pathologically diagnosed gastric cancer
3. Able to undergo radical resection (R0)
4. Scheduled for minimally invasive surgery (MIS)

Exclusion Criteria:

1. Pregnant or lactating women
2. Have received chemotherapy and radiation before surgery
3. Scheduled for open surgery
4. Subjects who do not understand or have not given informed consent
5. If healthcare provider (primary care physician) deems it difficult for you to exercise

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Shorts Physical Performance Battery(SPPB) | "1 day before surgery", "POD3", "POD 1month"
  SPPB is an objective measurement instrument of balance, lower extremity strength, and functional capacity. instrument of balance, lower extremity strength, and functional capacity. The test includes three different domains (walking, sit-to-stand and balance) to assess functional mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung-Il Kim, Principal Investigator — Department of Surgery, Yonsei University College of Medicine
Locations (1):
- Department of Surgery, Yonsei University College of Medicine, Seoul, South Korea